CLINICAL TRIAL: NCT00402701
Title: Pedestrian Behavior Following Implementation of a Walking School Bus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Baylor College of Medicine (Other); Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Brian Johnston, Professor: School of Medicine, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 04-3850-E/A
Record Dates: First submitted 2006-11-21; First posted 2006-11-22 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Obesity
Keywords: walking; motor activity; students; schools; transportation; motor vehicles
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Students in school with active walk-to-school promotion programs.
  Interventions: Behavioral: Walking School Bus Program
- 2 (No Intervention): Students in schools with access to standard school district transportation resources.

INTERVENTIONS:
Behavioral: Walking School Bus Program — Schoolwide promotion of walk to school. Facilitation of parent-led walking school bus routes.
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether a walking school bus program can increase the number of children walking to school and decrease the number of children driven by car to school.

DETAILED DESCRIPTION:
Walking to school is associated with higher levels of physical activity, which is an objective of Healthy People 2010. However, parents' concerns about safety have been identified as a barrier that prevents their children from walking to school. A walking school bus (WSB) addresses these concerns by providing a supervised period of physical activity on the way to school. A WSB is a group of children led to and from school by responsible adults who walk together along a set route. The peer-reviewed literature on active travel to school is sparse. We evaluated a WSB program, to test the hypothesis that it would increase the proportion of children walking and decrease the proportion of children driven by car to school.

Comparison: We conducted an 18-month controlled, quasi-experimental trial at three public elementary schools in Seattle, Washington. The intervention school was assigned a WSB coordinator who dedicated 10-15 hours/week establishing WSB routes and implementing school activities on pedestrian safety. Each "bus" had its own set route to school from different locations in the surrounding neighborhoods and was staffed by several parent leaders. The two control schools received standard Seattle Public Schools resources on walking to school including "Safe Route Maps," a traffic and safety committee, and school safety patrols. The primary outcomes were the proportions of children who walked with and without an adult or were driven by car to school. We used the test for independent proportions to compare the proportion of children transported to school at the intervention versus control schools.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in school
* Present on the day of the survey at one of 3 study schools.

Exclusion Criteria:

* Absent on the day of the survey at one of 3 study schools.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 735 (Actual)
Dates: Start 2004-11; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Proportion of children walking or driven by car to school at one-year | 1, 6 and 12 months post initiation of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Johnston, MD MPH, Principal Investigator — University of Washington
Locations (1):
- Harborview Injury Prevention Research Center - University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Mendoza JA, Levinger DD, Johnston BD. Pilot evaluation of a walking school bus program in a low-income, urban community. BMC Public Health. 2009 May 4;9:122. doi: 10.1186/1471-2458-9-122. PMID 19413910